CLINICAL TRIAL: NCT02595138
Title: Zoledronic Acid as Adjuvant Treatment of Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Ying Fan, Associate professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-039
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: zoledronic acid; triple-negative breast cancer; adjuvant treatment
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): zoledronic acid received
  Interventions: Drug: Zoledronic acid
- B (No Intervention): observation

INTERVENTIONS:
Drug: Zoledronic acid
  Arms: A

SUMMARY:
Triple-negative breast cancer is a special type of breast cancer with poor prgnosis and limited choices. Chemotherapy is the only choice of adjuvant systemic treatment options. Previous study suggested that zoledronic acid might have anti-tumor effect by eliminating the number of DTCs(Disseminated Tumor Cell )and had been proved to be effective as adjvant therapy in postmenopausal women whose breast cancer was Homonal receptor positive and who were receiving aromatase inhibitors. So it might be able to improve the survival of triple negative breast cancer patients.

DETAILED DESCRIPTION:
Triple negative breast cancer patients with high risk factor will be randomized to receive either zoledronic acid or observation after the completion of standard chemotherapy/radiotherapy. Recurrence status will be followed and Disease free survival will be compared. Overall survival is the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* •Adult women (≥ 18 years of age) with early stage breast cancer(stage II-III).

  * Histological confirmation of estrogen and/or progesterone-receptor negative (ER-), human epidermal growth factor receptor 2 negative (HER2 -) breast cancer.

ER/PR negative: nuclear reaction< 1%, HER2 negative: HER2; IHC 0,1+ or FISH/CISH (-) in case of IHC 2+

* axillary lymph node positive with other high risk factors: LVI, T>5CM, Grade III
* Patients finish standard chemotherapy and/or radiotherapy
* ECOG performance status of 0,1
* Adequate bone marrow, hepatic, and renal function
* Adequate bone marrow and coagulation function as shown by:
* Absolute neutrophil count (ANC) ≥ 1.5 109/L;Platelets>100 x109/L;Hemoglobin (Hgb) > 9.0g/dLINR < 2
* Adequate liver function as shown by:
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN
* Total serum bilirubin < 1.5 x ULN
* Adequate renal function as shown by:
* Serum creatinine< 1.5 x ULN
* Fasting serum cholesterol <300 mg/dL or 7.75 mmol/L and fasting triglycerides <2.5 x ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved.
* Written informed consent

Exclusion Criteria:

* •Another malignancy within 5 years prior to enrollment with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer.

  * Any severe and/or uncontrolled medical conditions, eg. currently active infection
  * Pregnant or lactating
  * Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years after last patient was enrolled
  the time from randomization to the time of disease progression or relapse or death

SECONDARY OUTCOMES:
overall survival | 5 years after last patient was enrolled
  the time from randomization to the time of death
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 28 days after last medication

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716